CLINICAL TRIAL: NCT00879450
Title: Evaluating the Impact of a New Complement to Physiotherapy Intervention for Positional Torticollis in Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical department where study was held was unable to continue collaboration
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Isabelle Gagnon, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PED-08-035
Record Dates: First submitted 2009-04-07; First posted 2009-04-10 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Torticollis
Keywords: Congenital muscular torticollis
MeSH Terms: conditions — Torticollis; Congenital torticollis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Booklet (Experimental)
  Interventions: Other: Booklet
- 2 standard (Active Comparator)
  Interventions: Other: Booklet

INTERVENTIONS:
Other: Booklet — booklet given to parents for home exercises

SUMMARY:
Children with a torticollis are usually referred for physiotherapy where they are evaluated, and given exercises as well as education to treat the condition. This study is being done in order to compare 2 methods of sharing information with parents of children with torticollis.

DETAILED DESCRIPTION:
160 children of less than 6 months of age will be recruited for the study and divided in 2 groups. Children of both groups will receive the same physiotherapy evaluation and exercises but parents will receive information handouts with one of two different types of illustrations and written instructions for home exercises.

ELIGIBILITY:
Inclusion Criteria:

* Aged newborn to 6 months at initial visit in physiotherapy,
* A diagnosis of PT made by a physician,
* At least 37 weeks of gestational age at delivery

Exclusion Criteria:

* Congenital muscular torticollis with fibrosis (confirmed diagnosis): because this is a rare condition that has a different rate of recovery,
* Presence of craniosynostosis (confirmed diagnosis made by a neurosurgeon),
* APGAR score of less than 7 at 5 minutes,
* Prescription of a Tubular Orthosis for Torticollis (TOT) collar or Botox intervention for the torticollis,
* Confirmed diagnosis of syndrome or neurological condition.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Neck range of motion measurements | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Children's Hospital, MUHC, Montreal, Quebec, Canada